CLINICAL TRIAL: NCT01642303
Title: The Effect of Vodcasting on Listening Comprehension
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nazila zarghi, faculty member, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Listening comprehension
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2010-01

CONDITIONS: Listen to Vodcast
Keywords: vodcasting,listening,language education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vodcasting (Experimental): students who listen to downloaded vodcasting
  Interventions: Other: vodcasting
- control (No Intervention): listen to the student book listening file
  Interventions: Other: no intervension

INTERVENTIONS:
Other: vodcasting — listening to downloaded vodcasting files
  Arms: vodcasting
Other: no intervension — Listen to student book listening files
  Arms: control

SUMMARY:
Improvement of the internet and its tremendous growth has caused significant progress in transformation of information. Nowadays in any place of the world and in any time of the day by accessing through internet every student can use different kinds of information in World Wide Web which let him to make the best decision what, how and when to study. One of these educational technologies which are beneficial to learners is vodcast or video recording which are accessible through the internet.This paper is going to examine the listening comprehension in EFL learners and whether it may be improved by using vodcasts. So106 language learners of four different classes of Iranian higher intermediate in an English institute were chosen for this study. These learners were pre-tested by IELTS Listening Comprehension. Two classes were chosen as subject group which consisted of 54 learners. The remaining two classes were chosen as control group which consisted of 52 learners. Both groups were taught Listening Impact book, but students in subject group were provided some vodcasts based on the topic of their lessons. After 12 weeks of teaching both groups were post-tested.listening comprehension will be compared using independent t-test and paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* EFL learner
* upper intermediate level

Exclusion Criteria:

* Other levels

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
improving listening comprehension | up to 12 weeks
  The outcome mesures will be completed up to 12 weeks using IELTS listening comprehension tests